CLINICAL TRIAL: NCT00516984
Title: Osteopathic Manipulative Treatment and Its Relationship to Autonomic Nervous System Activity as Demonstrated by Heart Rate Variability
Brief Title: Osteopathic Manipulative Treatment and Its Relationship to Autonomic Nervous System Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Charles Henley, DO, MPH, OU Health Sciences Center - Tulsa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUIRB 12024
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Relationship between Osteopathic Manipulative Therapy (OMT) and the autonomic nervous system; LF/HF ratio
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): No-touch control condition applied while subject was at a 50-degree head-up tilt.
  Interventions: Procedure: Placebo
- Sham (Sham Comparator): Touch-only sham treatment applied while subject was at a 50-degree head-up tilt.
  Interventions: Procedure: Sham
- OMT (Active Comparator): Cervical myofascial OMT applied while subject was at a 50-degree head-up tilt.
  Interventions: Procedure: OMT

INTERVENTIONS:
Procedure: Placebo — No-touch control condition applied while subject was at a 50-degree head-up tilt.
  Arms: Placebo
Procedure: Sham — Touch-only sham treatment applied while subject was at a 50-degree head-up tilt.
  Arms: Sham
Procedure: OMT — Cervical myofascial OMT applied while subject was at a 50-degree head-up tilt.
  Arms: OMT

SUMMARY:
The relationship between Osteopathic Manipulative Therapy (OMT) and the autonomic nervous system is poorly understood. This study quantifies that relationship and demonstrates a cause and effect. It is hypothesized that cervical myofascial release increases vagal tone.

DETAILED DESCRIPTION:
For most osteopathic physicians the validation of osteopathic manipulative treatment (OMT) has been largely observational and based on patient outcomes such as improvement in pain scales, range of motion, and other empiric measures.1,2 However, the osteopathic profession has long recognized a relationship between the autonomic nervous system and the function of the body in health and disease, although there is relatively little quantitative data evaluating the relationship between manipulation and the autonomic nervous system.3,4

A theoretical basis for the action of OMT and its effect in the body has been advanced based on autonomic activation causing concomitant vasodilatation, smooth muscle relaxation, and increased blood flow, resulting in improved range of motion, decrease in pain perception, or change in tissue. Until recently this association remained largely a theoretical consideration due to the inability to accurately measure autonomic activity directly. Over the past two decades indirect methods have been developed and refined to provide noninvasive markers of autonomic balance,5,6 with heart rate variability (HRV) being commonly used. HRV is based on the inherent variation of the R-to-R intervals of a standard electrocardiogram (ECG), with these variations largely due to changes in autonomic balance at the sinus node.6-8

Spectral analysis of heart rate variability has been used to study autonomic balance in humans, and it is generally accepted that the high frequency (HF) component (0.15-0.4 Hz) can be used as a marker for vagal modulation of heart rate. Although it is tempting to use the low frequency (LF) component (0.04-0.15 Hz) as a marker for sympathetic activity, its specificity is less clear. Pagani and colleagues9,10 have hypothesized that when the LF component is expressed in normalized units (LFnu) it becomes a better marker of sympathetic modulation of heart rate. For most studies using spectral analysis, the LF/HF ratio is used and considered by many to be a good index of sympathovagal balance.6,7,9,10

The confidence given to the LF/HF ratio accurately reflecting autonomic balance is significantly influenced by experimental design. A tilt protocol involving postural change from horizontal to upright can be used to calibrate the change in the LF/HF ratio which occurs between the two positions and thus set a physiological range for sympathetic and vagal modulation of heart rate. An experimental procedure then can be implemented where comparisons are made of the changes in the LF/HF ratios that occur when the body is shifted from the horizontal to the upright position under conditions with application of an intervention versus without the intervention. In this manner, an experimentally mediated change in LF/HF ratio (i.e., with intervention) can be calibrated against a physiologically relevant change in ratio (i.e., without intervention).

This approach was used by these investigators in a pilot study (n=9 healthy, adult volunteers, 3 females and 6 males) which showed that the LF/HF ratio changed from a mean of 1.75+1.40 (mean+SD) in the horizontal position to a mean of 6.00+1.20 in the 50-degree head-up position. This change reflects an increase in sympathetic tone. Mean heart rate in these subjects increased from 61+7 bpm to 78+2 bpm in the head-up position. The subjects then were treated in the 50-degree head-up position with an OMT procedure, cervical myofascial release, which is thought to increase vagal tone. After the procedure was applied, the LF/HF ratio decreased back down to 1.75+1.58, even though the subjects were still in the head-up position. These data support the initial hypothesis that specific OMT procedures can modulate vagal tone, and also provide information relating to the significance of the LF/HF change. That is, the application of OMT reversed the increase in the ratio that occurs in the 50-degree head-up position.

We conducted a continuation project to further examine the association between OMT and autonomic nervous system activity as demonstrated by HRV, studying the hypothesis that cervical myofascial release increased vagal tone. In a within subjects (repeated measures) design, we examined the effect of OMT on HRV in comparison with sham treatment (touch only) and control (no touch) conditions.

ELIGIBILITY:
Inclusion Criteria:

Twenty-eight (28) study subjects then were selected by their response to a general questionnaire, which indicated suitability for the study, and assessed by the following inclusion criteria:

* written informed consent
* normal healthy adults older than 19 years and younger than 50 years
* normal ECG
* normal blood pressure based on criteria published in the Seventh Report of the U.S. Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC-7).

Exclusion Criteria:

* Exclusion criteria included chronic cardiovascular disease (heart failure, myocardial infarction, or hypertension)
* diabetes
* asthma
* pregnancy
* smoking
* premature ventricular contractions exceeding 20% of total heart beats
* resting supine heart rate greater than 75 bpm or less than 45 bpm, systolic blood pressure greater than 140 mmHg or less than 90 mmHg
* failure of heart rate to increase with passive tilt (50-degrees head-up)
* Long-distance runners and other conditioned athletes also were excluded

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Normalized low frequency and high frequency components of HRV, including LF/HF ratio. Comparisons between measurements taken at a 50-degree tilt with those taken at pre- and post-intervention in the horizontal position. | Treatments administered in separate sessions at least 24 hours apart.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Henley, D.O., MPH, Principal Investigator — OUHSC; Frances Wen, Ph.D., Principal Investigator — OUHSC; Bruce Benjamin, Ph.D., Principal Investigator — OSU; Douglas Ivins, M.D., Principal Investigator — OUHSC; Miriam Mills, M.D., Principal Investigator — OSU
Locations (1):
- OSU, Tulsa, Oklahoma, United States

REFERENCES:
- [Derived] Henley CE, Ivins D, Mills M, Wen FK, Benjamin BA. Osteopathic manipulative treatment and its relationship to autonomic nervous system activity as demonstrated by heart rate variability: a repeated measures study. Osteopath Med Prim Care. 2008 Jun 5;2:7. doi: 10.1186/1750-4732-2-7. PMID 18534024